CLINICAL TRIAL: NCT06087796
Title: Topical Pentoxifylline; Metformin Versus Betamethasone in the Treatment of Alopecia Areata: a Clinical and Dermoscopic Study.
Brief Title: Topical Pentoxifylline; Metformin Versus Betamethasone in the Treatment of Alopecia Areata.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Khaled Mohamed Mostafa, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Topicals in Alopecia areata
Record Dates: First submitted 2023-09-24; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Alopecia Areata
Keywords: metformin; pentoxiphylline; betamethasone valerate; alopecia areata
MeSH Terms: conditions — Alopecia Areata | interventions — Betamethasone Valerate; Betamethasone; Pentoxifylline; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical betamethasone (Active Comparator): Group A will include 20 patients and will receive topical betamethasone valerate 0.1% cream.
  Treatment will be applied twice daily for 6 months or until complete resolution, whichever is sooner.
  Interventions: Drug: Betamethasone Valerate 0.1% Cream
- Topical pentoxifylline (Experimental): Group B will include 20 patients who will receive topical pentoxifylline 2% gel.
  Treatment will be applied twice daily for 6 months or until complete resolution, whichever is sooner.
  Interventions: Drug: Pentoxifylline
- Topical metformin (Experimental): Group C will include 20 patients who will receive topical metformin 10% gel. Treatment will be applied twice daily for 6 months or until complete resolution, whichever is sooner.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Betamethasone Valerate 0.1% Cream — Topical treatment modality for alopecia areata.
  Other Names: Topical betamethasone
  Arms: Topical betamethasone
Drug: Pentoxifylline — Topical treatment modality for alopecia areata.
  Other Names: topical pentoxifylline
  Arms: Topical pentoxifylline
Drug: Metformin — Topical treatment modality for alopecia areata.
  Other Names: Topical metformin
  Arms: Topical metformin

SUMMARY:
To compare the efficacy and safety of topical pentoxifylline 2% gel and topical metformin 10% gel versus topical betamethasone valerate 0.1% cream, in treatment of patchy alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a common tissue-specific autoimmune disease characterized by non-scaring hairloss.

Alopecia areata affects around 2.1% of the population at a point of their life. It affects both males and females without significant difference. Alopecia areata can occur at any age with a peak incidence in the twenties and thirties, however, the younger the attack, the more severe the course of the disease.

Alopecia areata is subdivided into 3 subgroups depending on the extent and site of hair loss; these are patchy alopecia areata, alopecia totalis and alopecia universalis. The most common presentation is patchy alopecia areata which presents as a rounded or oval patch(es) of hairloss.

Dermoscopy is a noninvasive tool which aids the diagnosis of alopecia areata. Characteristic dermoscopic features in AA include black dots (BDs), yellow dots (YDs), exclamation mark hairs (EHs), and broken hairs (BHs). BDs and EHs are the most specific findings in AA and correlate with disease activity, whereas YDs are seen in all the stages of the disease and correlate with disease severity.

The course of AA is unpredictable, with spontaneous remission during the first 6-12 months occurs in 30-50% of patients.

It has been hypothesized to be a T-cell mediated immune response disease through CD4+ and CD8+ that violate the immune privilege of the anagen hair follicle, leading to loss of the growing hair shaft (Islam et al., 2015). Studies regarding the pathogenesis of AA reveal an intricate complexity involving multiple factors including immunology, genetics, the environment, and potentially the microbiome.

Furthermore, it can be associated with other autoimmune diseases such as thyroid disease, diabetes mellitus type 2, vitiligo, systemic lupus erythematosus, psoriasis, inflammatory bowel disease and rheumatoid arthritis.

Alopecia areata has a major impact on patient's quality of life as it affects patient's self-esteem and his social relationships. Moreover, it was found to be associated with different psychiatric disorders such as depression and generalized anxiety disorder; which explains the need for early and appropriate treatment for alopecia areata.

There are many treatment modalities for AA including topical treatment, intralesional injections, systemic corticosteroids, systemic immunosuppressant like methotrexate or cyclosporine, excimer laser and photochemotherapy. Recently there's an emergence of new treatments for AA such as; Janus kinases signal transducer and activator of transcription proteins (JAK-STAT) inhibitors (baricitinib, ritlecitinib, deuruxolitinib, brepocitinib) as a promising new class of agents that can induce significant hair regrowth, phosphodiesterase-4 inhibitors (apremilast) and the biologics (dupilumab, secukinumab and aldesleukin) appear to have limited efficacy so far. However, there's no uniformly effective medication for this disease.

In the last few years, several topical agents were suggested as possible therapeutic options for patchy AA such as topical methotrexate and topical calcipotriol.

Topical corticosteroids are frequently used in treatment of patchy alopecia areata, potent and moderately potent steroids are the first line treatment in children and adults who can't tolerate intralesional steroid injection in patchy alopecia areata. However, they have a low success rate in treatment of alopecia totalis and universalis.

They have various formulations (foams, creams, lotions, ointment and solution) that can be used and have fewer side effects than systemic therapy.

Corticosteroids are known to have a strong inhibitory effect on activation of T-lymphocytes providing that AA is a T-cell mediated autoimmune response thus decreasing the inflammation around hair bulb region, allowing hair follicles to enter a normal hair cycle.

Side effects of topical formulations of corticosteroids include; folliculitis, that is the most common, post-inflammatory hyper/hypopigmentation, atrophy, and telangiectasia.

Pentoxifylline (PTX) is a methylxanthine derivative, which acts as a phosphodiesterase inhibitor and it is primarily used in microcirculatory disorders. Pentoxifylline also has an immunomodulatory effect through inhibition of several cytokines including TNF -α, IL-1, and IL-6 that play a role in inflammation. It has also been shown to suppress B cells, T cells, and neutrophils as well as decrease the expression of endothelial adhesion molecules.

Oral PTX has been used in dermatological disorders such as alopecia areata with beneficial effects. To the best of our knowledge there is no previous study reported the use of topical PTX in treatment of AA, however, there is only one study that used intralesional PTX in treatment of patchy AA. In this study intralesional PTX was tried both alone and in combination with intralesional triamcinolone acetonide (TRA) versus intralesional triamcinolone acetonide alone. This study found that the combined drug usage (TRA & PTX) had the best results followed by PTX alone and then triamcinolone acetonide alone (72.0%, 60.0%, and 32.0%, respectively).

Metformin is commonly used as a first-line treatment for type 2 diabetes. It reduces glucose levels by improving peripheral tissues' sensitivity to insulin, decreasing the liver's gluconeogenesis and reducing intestinal glucose absorption. Recently, several studies reported the usefulness of metformin in treatment of different autoimmune disorders such as scleroderma and systemic lupus erythematosus due to its immunomodulatory actions, as a new deal of an old drug.

Metformin can modulate the immune system by increasing the cellular AMP-activated protein kinase (AMPK) enzyme that inhibits the Janus kinase/signal transducers and activators of transcription (JAK-STAT) and mammalian target of Rapamycin (mTOR) intracellular signaling pathways. Inhibition of the mTOR pathway prevents the proliferation and differentiation of T lymphocytes into cytotoxic T cells, which are the leading causes of hair follicle destruction in AA. It also promotes the proliferation of regulatory T cells (Tregs); that play a crucial role in maintaining the immune privilege of hair follicles as they produce transforming growth factor-1 (TGF-1) that contributes to maintaining immune privilege.

Inhibition of the JAK-STAT pathway by metformin prevents the production of cytokines, including interferon gamma (IFN-γ) and interleukin 17 (IL-17). The production of these cytokines is necessary to collapse the immune privilege status of the hair follicle. Moreover, metformin was found to enhance the proliferation and differentiation of hair follicle stem cells, aiding hair follicle regeneration.

Oral metformin has been used in different dermatological diseases such as hormonal acne, hidradenitis suppurativa (HS) and acanthosis nigricans in which it may act through improving hyperinsulinemia. Additionally, it was found effective when used topically in treatment of melasma with an equivalent effect to triple combination cream (TCC), and acne vulgaris.

Interestingly, topical metformin was reported to be successful in treating central centrifugal Cicatricial alopecia in a single case report.

Recently, Kokhabi et al., 2023 hypothesized that topical metformin may be effective in AA due to its anti-inflammatory and immunomodulatory actions, however, to the best of our knowledge, no clinical trials have been conducted yet and such a hypothesis still needs to be proven by future studies.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of patchy alopecia areata of scalp involving < 50% of the total scalp confirmed by dermoscopy of both males and females.
* patients age between 6 and 60 years old.

Exclusion Criteria:

* Alopecia totalis and alopecia universalis.
* Cicatricial alopecia.
* Other causes of hair loss such as; endocrine or immunological disease.
* Skin disease in the affected area.
* Hypersensitivity or allergy to any of the treatment products used.
* Patient using treatment (topical or systemic) for alopecia areata in the last 2 months.
* Systemic administration of any of the three test drugs (pentoxifylline, metformin and steroids).
* Pregnant and lactating females.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of hair regrowth in alopecia areata using SALT score. | 8 months
  The scalp is divided into four parts on the basis of surface area as follows: vertex or top = 40% (0.40), right side = 18% (0.18), left side = 18% (0.18) and the posterior aspect = 24% (0.24). Percentage of hair loss in any of the four areas is multiplied by the percentage of the scalp covered in that area. The SALT score is the sum of the percentage of hair loss in all the areas mentioned above.

CONTACTS AND LOCATIONS:
Overall Officials: Nada K. Mostafa, bachelor, Principal Investigator — Assuit university hospital
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirzoyev SA, Schrum AG, Davis MDP, Torgerson RR. Lifetime incidence risk of alopecia areata estimated at 2.1% by Rochester Epidemiology Project, 1990-2009. J Invest Dermatol. 2014 Apr;134(4):1141-1142. doi: 10.1038/jid.2013.464. Epub 2013 Nov 11. No abstract available. PMID 24202232
- [Background] Islam N, Leung PS, Huntley AC, Gershwin ME. The autoimmune basis of alopecia areata: a comprehensive review. Autoimmun Rev. 2015 Feb;14(2):81-9. doi: 10.1016/j.autrev.2014.10.014. Epub 2014 Oct 12. PMID 25315746
- [Background] Juarez-Rendon KJ, Rivera Sanchez G, Reyes-Lopez MA, Garcia-Ortiz JE, Bocanegra-Garcia V, Guardiola-Avila I, Altamirano-Garcia ML. Alopecia Areata. Current situation and perspectives. Arch Argent Pediatr. 2017 Dec 1;115(6):e404-e411. doi: 10.5546/aap.2017.eng.e404. English, Spanish. PMID 29087123
- [Background] Karimkhani C, Boyers LN, Prescott L, Welch V, Delamere FM, Nasser M, Zaveri A, Hay RJ, Vos T, Murray CJ, Margolis DJ, Hilton J, MacLehose H, Williams HC, Dellavalle RP. Global burden of skin disease as reflected in Cochrane Database of Systematic Reviews. JAMA Dermatol. 2014 Sep;150(9):945-51. doi: 10.1001/jamadermatol.2014.709. PMID 24807687
- [Background] Zargari O. Pentoxifylline: a drug with wide spectrum applications in dermatology. Dermatol Online J. 2008 Nov 15;14(11):2. PMID 19094840
- [Background] Speirs C, Williams JJL, Riches K, Salt IP, Palmer TM. Linking energy sensing to suppression of JAK-STAT signalling: A potential route for repurposing AMPK activators? Pharmacol Res. 2018 Feb;128:88-100. doi: 10.1016/j.phrs.2017.10.001. Epub 2017 Oct 13. PMID 29037480
- [Background] Speiser JJ, Mondo D, Mehta V, Marcial SA, Kini A, Hutchens KA. Regulatory T-cells in alopecia areata. J Cutan Pathol. 2019 Sep;46(9):653-658. doi: 10.1111/cup.13479. Epub 2019 May 15. PMID 30989699
- [Background] Araoye EF, Thomas JAL, Aguh CU. Hair regrowth in 2 patients with recalcitrant central centrifugal cicatricial alopecia after use of topical metformin. JAAD Case Rep. 2020 Jan 22;6(2):106-108. doi: 10.1016/j.jdcr.2019.12.008. eCollection 2020 Feb. No abstract available. PMID 32016152
- [Background] Tawfeek HM, Abou-Taleb DAE, Badary DM, Ibrahim M, Abdellatif AAH. Pharmaceutical, clinical, and immunohistochemical studies of metformin hydrochloride topical hydrogel for wound healing application. Arch Dermatol Res. 2020 Mar;312(2):113-121. doi: 10.1007/s00403-019-01982-1. Epub 2019 Oct 16. PMID 31620870
- [Background] Jha AK, Udayan UK, Roy PK, Amar AKJ, Chaudhary RKP. Dermoscopy of alopecia areata-a retrospective analysis. Dermatol Pract Concept. 2017 Apr 30;7(2):53-57. doi: 10.5826/dpc.0702a12. eCollection 2017 Apr. PMID 28515996
- [Result] El-Taweel AI, Akl EM. Intralesional pentoxifylline injection in localized alopecia areata. J Cosmet Dermatol. 2019 Apr;18(2):602-607. doi: 10.1111/jocd.12796. Epub 2018 Oct 9. PMID 30302901